CLINICAL TRIAL: NCT02203552
Title: Randomized Placebo Controlled Study of Minocycline for Amelioration of Chemotherapy Induced Affective Disorders
Brief Title: Minocycline Hydrochloride in Reducing Chemotherapy Induced Depression and Anxiety in Patients With Stage I-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-13165; NCI-2014-00851 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Anxiety Disorder; Depression; Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Breast Neoplasms | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (minocycline hydrochloride) (Experimental): Beginning 1 week prior to chemotherapy, patients receive minocycline hydrochloride orally PO BID for 9 weeks. Laboratory biomarker analysis will also be obtained weekly on protocol. Questionnaire administration weekly.
  Interventions: Drug: minocycline hydrochloride; Other: laboratory biomarker analysis; Other: Questionnaire administration
- Arm II (placebo) (Placebo Comparator): Beginning 1 week prior to chemotherapy, patients receive placebo PO BID for 9 weeks. Laboratory biomarker analysis will also be obtained weekly on protocol. Questionnaire administration weekly.
  Interventions: Other: placebo; Other: laboratory biomarker analysis; Other: Questionnaire administration

INTERVENTIONS:
Drug: minocycline hydrochloride — 100 mg bid given by mouth for 9 weeks
  Other Names: Dynacin; Minocin; Minomax; Minomycin
  Arms: Arm I (minocycline hydrochloride)
Other: placebo — Placebo given by mouth for 9 weeks
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative blood levels for cortisol, high sensitivity c-reactive protein (hs-CRP) and inflammatory factors including but not limited to IL-6, TNF-α, IL-1β, and MCP-1 will also be obtained weekly on protocol.
  Other Names: special studies; Correlative studies
Other: Questionnaire administration — The CES-D and STAI will be administrated weekly.
  Other Names: Ancillary studies

SUMMARY:
This randomized clinical trial studies how well minocycline hydrochloride works in reducing chemotherapy induced depression and anxiety in patients with stage I-III breast cancer. Minocycline hydrochloride may prevent changes in memory and thinking and improve the quality of life of breast cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate anxiety and depression in women with stages I-III breast cancer during the first 8 weeks of doxorubicin-based adjuvant therapy randomized to receive either minocycline (minocycline hydrochloride) or placebo.

II. To evaluate markers of neuro-inflammation as assessed by blood based inflammatory cytokines and C11-choline positron emission tomography (PET) in women with stages I-III breast cancer during the first 8 weeks of doxorubicin-based adjuvant therapy randomized to receive either minocycline or placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Beginning 1 week prior to chemotherapy, patients receive minocycline hydrochloride orally (PO) twice daily (BID) for 9 weeks.

ARM II: Beginning 1 week prior to chemotherapy, patients receive placebo PO BID for 9 weeks.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer stages I-III initiating first line adjuvant or neoadjuvant doxorubicin hydrochloride (DOX) chemotherapy
* Postmenopausal defined as amenorrhea > 12 months or follicle stimulating hormone (FSH) and estradiol in institutional postmenopausal range
* Ability to understand English and read and write at the 8th grade level and give a written informed consent document
* For additional cohort, women with breast cancer stages I-III who currently on or within 18 months of completing first line adjuvant or neoadjuvant DOX chemotherapy or other chemotherapy for breast cancer.

Exclusion Criteria:

* Rheumatoid arthritis and other types of autoimmune and inflammatory joint disease, with the exception of osteoarthritis and fibromyalgia
* Concurrent other malignancy or metastatic malignancy of any kind
* Reported diagnosis of major depression or anxiety disorder prior to breast cancer (BC) diagnosis
* Currently prescribed psychotropic medications including anti-depressants
* Known bleeding disorders
* History of diabetes mellitus, heart disease or stroke
* Current use of warfarin or other anticoagulants
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, hypertension, or psychiatric illness/social situation that would limit compliance with study requirements
* Pregnant or nursing women
* Concurrent use of daily full dose aspirin (>= 325 mg/day), nonsteroidal anti-inflammatory drugs (NSAIDs) or NSAID-containing products or steroids; one month washout period is required prior to randomization
* Unable to give informed consent
* Tetracycline allergy
* Any contraindication to magnetic resonance imaging (MRI)/PET examination including but not limited to ferromagnetic metal in the body, pacemaker, or severe claustrophobia; (however, this portion is optional and if patient is otherwise eligible, can enroll in study without participating in imaging study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvaneswari Ramaswamy, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from June 2015 until June 2020
Period: Overall Study
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo) | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.0) | 52.7 (11.8) | 51.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Changes in Center for Epidemiological Studies Depression Scale (CES-D) Scores
Description: CES-D scale a short self-reported scaled designed to measure depressive symptomology in the general population. At baseline, depressive symptom severity will be assessed using the CES-D instrument. Evaluation of the patients assessment if suicidal ideation is reported at baseline. A value of 0, 1, 2, or 3 is assigned to a response depending upon positively or negatively. The subject will be withdrawn from the administrated serially every cycle starts on protocol during clinic visits (Patients will self-administer forms given out by research coordinator).The internal consistency for the STAI is .95; higher scores indicate greater anxiety.41 The internal consistency for the CES-D is approximately .85 among BC patients,42 and an important benefit of using this scale in medical studies is that it is relatively unaffected by physical symptoms. Total scores range from 0-60 with higher scores reflecting greater depressive symptoms. The 95% confidence intervals of the depression change from b
Time Frame: Baseline to 9 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 28 | 28
score on a scale | 0.57 [-2.87 to 4] | -3.18 [-6.4 to 0.03]

2. Primary Outcome: Changes in the State Trait Anxiety Index (STAI) Scores
Description: The mean changes over time in State Trait Anxiety Index (STAI) scores from baseline to the end of study for the two study groups. The influences of covariate, such as disease stage and depression drug usage, will be considered in the mixed models as exploratory analyses. The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).The 95% confidence intervals of the change in the primary outcome measures from baseline to the end of study and the differences between the treatment and placebo groups will be estimated based on the models.
Time Frame: Baseline to 9 weeks
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 28 | 28
scores on a scale | -5.86 [-11.69 to -0.04] | -9.41 [-16.38 to -2.44]

3. Secondary Outcome: Changes in Hamilton Anxiety Rating Scale Scores
Description: The 95% confidence intervals of the anxiety change from baseline to the end of study and the difference between the treatment and placebo groups. The influences of covariate, such as disease stage and depression drug usage, will be considered in the mixed models as exploratory analyses. In addition, change overtime of all outcomes for each individual will be plotted to visually explore any patterns and to generate hypothesis to be tested in future studies.
Time Frame: Baseline to 9 weeks
Population: Data was not collected and analyzed
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Changes in Hamilton Rating Scale for Depression Scores
Description: The 95% confidence intervals of the depression change from baseline to the end of study and the difference between the treatment and placebo groups. The influences of covariate, such as disease stage and depression drug usage, will be considered in the mixed models as exploratory analyses. In addition, change overtime of all outcomes for each individual will be plotted to visually explore any patterns and to generate hypothesis to be tested in future studies.
Time Frame: Baseline to 9 weeks
Population: Data not collected or analyzed
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Changes in Inflammatory Blood Markers
Description: Scatter plots will be used to explore the pair-wise correlation among the changes of CES-D and STAI scores, blood biomarkers changes, and PET/MRI measures. A statistical model will be used to explore whether the blood based biomarkers and PET/MRI measures can be used to predict the changes in CES-D and STAI scores, which then could be used as potential surrogate markers in future studies.
Time Frame: Baseline to 6 months
Measure: Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 28 | 28
pg/ml
  IL-1b | 0.04 [-0.2 to 0.29] | 0 [-0.13 to 0.12]
  IL-6 | 0.17 [0.05 to 0.39] | 0.26 [0.12 to 0.41]
  IL-8 | 0.07 [-0.04 to 0.19] | 0.14 [0.01 to 0.27]
  TNF-a | 0.18 [0.05 to 0.32] | 0.11 [-0.01 to 0.22]
  TNF-RII | 0.11 [0.04 to 0.17] | 0.06 [0.02 to 0.1]

6. Secondary Outcome: Changes in the PET/MRI Measures
Description: as for outcome 5
Time Frame: Baseline to 6 months
Population: Data not collected and analyzed
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Toxicity will be monitored from the beginning of the study through study follow-up, an average of 1 year.
Description: Toxicity will be monitored during study visits and telephone calls using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 (CTCAE) of the National Cancer Institute will be used Grade 3, 4 and 5 toxicities will be reported as adverse events.
Arm/Group | Arm I (Minocycline Hydrochloride) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 28/28 | 28/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Minocycline Hydrochloride) (N=28) | Arm II (Placebo) (N=28)
Hypertension (Vascular disorders) | 28 (28) | 28 (28)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (22) | 21 (21)
Anemia (Blood and lymphatic system disorders) | 28 (28) | 28 (28)
Fatigue (General disorders) | 18 (18) | 22 (22)
Nausea (Gastrointestinal disorders) | 18 (18) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 8 (8) | 9 (9)
Anxiety (Psychiatric disorders) | 10 (10) | 13 (13)
Headache (Nervous system disorders) | 11 (11) | 14 (14)
Mucositis (Gastrointestinal disorders) | 8 (8) | 13 (13)
Constipation (Gastrointestinal disorders) | 10 (10) | 10 (10)
Dizziness (Nervous system disorders) | 11 (11) | 10 (10)
Vomiting (Gastrointestinal disorders) | 7 (7) | 12 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (11)
Pain (General disorders) | 11 (11) | 7 (7)
Bone Pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6)
Edema Limbs (General disorders) | 5 (5) | 12 (12)
Peripheral motor neuropathy (Nervous system disorders) | 9 (9) | 8 (8)
Depression (Psychiatric disorders) | 6 (6) | 7 (7)
Insomnia (Psychiatric disorders) | 7 (7) | 8 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Hot Flashes (Vascular disorders) | 6 (6) | 5 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Epistaxis (Gastrointestinal disorders) | 4 (4) | 4 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 4 (4) | 3 (3)
Fever (General disorders) | 4 (4) | 3 (3)
Platelet count decreased (Investigations) | 2 (2) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 5 (5)
Hypothyroidism (Immune system disorders) | 0 (0) | 6 (6)
Paresthesia (Nervous system disorders) | 5 (5) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 5 (5)
Arthritis (Immune system disorders) | 1 (1) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Eye disorders (Eye disorders) | 1 (1) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT02203552/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT02203552/ICF_001.pdf